CLINICAL TRIAL: NCT04315428
Title: Study of Swaddling on Tactile Learning in Premature Infants
Acronym: EMMASENS
Status: Completed | Type: Observational
Sponsor: University Hospital, Grenoble (Other)
Collaborators: GeneveUniversity (Unknown)
Responsible Party: Sponsor
Other Study IDs: 38RC18.060
Record Dates: First submitted 2019-12-19; First posted 2020-03-19 (Actual); Last update posted 2020-03-19 (Actual); Status verified 2020-03

CONDITIONS: Premature Newborn
MeSH Terms: conditions — Premature Birth

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 2 Years
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- premature swaddled: the childs in this group will be wrap in a lange (swaddled)
  Interventions: Behavioral: swaddling
- premature no swaddled: the childs in this group will be not swaddled
  Interventions: Behavioral: no swaddling

INTERVENTIONS:
Behavioral: swaddling — The two experimenters together evaluate the child's state of awakening throughout the experiment. If the child is considered by both experimenters to be too restless or too sleepy, the experiment is immediately stopped and postponed
  Groups: premature swaddled
Behavioral: no swaddling — The two experimenters together evaluate the child's state of awakening throughout the experiment. If the child is considered by both experimenters to be too restless or too sleepy, the experiment is immediately stopped and postponed
  Groups: premature no swaddled

SUMMARY:
Explore the sensorially of the premature newborn that is fundamental to adapting the care environment to these hospitalized babies

DETAILED DESCRIPTION:
Indeed, the challenge is to offer them an environment adapted to their sensory skills, so as not to alter their development.

This is in line with the customized care development, better known as the Anglo-Saxon term of Neonatal Individualised Developmental Care and Assessment Program.

The aim is thus to promote later the cognitive development of these children

ELIGIBILITY:
Inclusion Criteria:

* Children born prematurely and aged 28 to 35 Weeks of Amenorrhoea, regardless of their postnatal age

Exclusion Criteria:

premature newborns with

* associated anomalies syndrome
* abnormal cranial ultrasonography with stage III or IV intraventricular hemorrhage or periventricular cavitary leukaemia
* those receiving sedative or convulsive treatment during the experiment
* those whose grasping reflex is absent

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: Children born prematurely and hospitalized in the neonatal and neonatal resuscitation unit at the University Hospital of Grenoble
Sampling Method: Non-Probability Sample
Enrollment: 40 (Actual)
Dates: Start 2018-12-12 (Actual); Primary Completion 2019-05-23 (Actual); Study Completion 2019-05-23 (Actual)

PRIMARY OUTCOMES:
time required to habituate a first object (corresponding to a time when the object is held repeatedly) and time required to present a new object (corresponding to the property of discrimination) | up to 3 months max
  time required to habituate a first object (corresponding to a time when the object is held repeatedly) and time required to present a new object (corresponding to the property of discrimination)

SECONDARY OUTCOMES:
Compare cognitive development at 2 years in both groups | between first evaluation and 2 years
  Global development quotient, derived from the Brunet-Lezine scale, (performed systematically as part of the normal follow-up of premature babies in the N&D care network).
  the Brunet-Lezine scale : it is a global development quotient (QD) which is calculated and which corresponds to a standardized score (average of 100). Higher score corresponds to better child development

CONTACTS AND LOCATIONS:
Overall Officials: Leïla MARCUS, Dr, Principal Investigator — University Hospital, Grenoble
Locations (1):
- Chu Grenoble Alpes, Grenoble, France

REFERENCES:
- [Derived] Lejeune F, Delacroix E, Gentaz E, Berne-Audeoud F, Marcus L, Debillon T. Influence of swaddling on tactile manual learning in preterm infants. Early Hum Dev. 2021 Feb;153:105288. doi: 10.1016/j.earlhumdev.2020.105288. Epub 2020 Dec 3. PMID 33291020